CLINICAL TRIAL: NCT03596346
Title: Evaluation of Safety and Tolerability of a Rapeseed Food Ingredient Among Generally Healthy Consumers - A Randomized Double-blind, Controlled Parallel-group Four-week Intervention Trial
Brief Title: Evaluation of Safety and Tolerability of a Rapeseed Food Ingredient
Acronym: RYPSI-ING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avena Nordic Grain Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MFAV009
Record Dates: First submitted 2018-06-19; First posted 2018-07-23 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-06

CONDITIONS: Food Safety
Keywords: Rapeseed; Ingredient; Safety; Tolerability
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Active Comparator): 20 g of rapeseed ingredient (RI) daily
  Interventions: Other: Rapeseed ingredient (RI)
- Control group (Placebo Comparator): 0 g of rapeseed ingredient (RI) daily
  Interventions: Other: Control product without added RI

INTERVENTIONS:
Other: Rapeseed ingredient (RI) — 2 snack bars daily containing 10 g of RI each.
  Arms: Test group
Other: Control product without added RI — 2 snack bars daily containing 0 g of RI.
  Arms: Control group

SUMMARY:
The study is designed to assess the safety and tolerability of a novel food ingredient produced from rape seeds supplied as a snack-bar in a 4-week controlled intervention.

DETAILED DESCRIPTION:
An 4-week randomized, double-blind, controlled, parallel-group intervention for assessment of safety and tolerability of a novel rape seed ingredient (RI) followed by a 2-week follow-up period. Baseline measures for digestive symptom frequency questionnaire (DSFQ), blood safety tests and body mass index (BMI) will be collected at screening visit. At the randomization visit, participants' eligibility will be confirmed, and they will be randomly allocated into 2 parallel groups consuming either 20 g (test group) or 0 g (control group) of RI within 2 daily snack bars. During the intervention and follow-up periods participants will bi-weekly respond to a GI symptom questionnaire including DSFQ, stool frequency and stool consistency, and palatability items. At the end of the intervention period (week 4) a clinic visit including BMI and AE recording and blood safety tests will be held.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age 18-75 years (inclusive)
* Body mass index (BMI) 18.5 - 30 (inclusive)
* Good general health according to medical history and current health status

Exclusion Criteria:

* Allergy or sensitivity to any ingredient of the study products
* Nut or mustard allergy
* Any major diseases or malfunctions including i. Inflammatory bowel disease or functional bowel disorder or any major gastrointestinal medical condition ii. type 1 or 2 diabetes requiring medication iii. active hepatic, kidney or thyroid disease or disorder except if subject on thyroid replacement therapy iv. myocardial infarction, unstable symptomatic angina pectoris, or transient ischemic attack or stroke within 3 months prior to screening v. cancer or cancer treatment within 5 years prior to screening (not including basal cell carcinoma)
* Medication used for treatment of elevated blood glucose levels
* Pregnancy, lactation or planned pregnancy during the trial
* Clinically significant abnormalities in safety laboratory values according to the investigator
* Strict low-carbohydrate or low-fat diet
* Participation in another clinical trial in the preceding 1 month
* Likelihood of any health or safety risk according to the Investigator
* Likelihood of non-compliance according to the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Change in digestive symptom frequency score | Change from week 0 to week 4
  Change in composite frequency score of four gastrointestinal (GI) symptoms according to the digestive symptom frequency questionnaire (DSFQ; combined score for four questions ranging from 0 to 16; subjective evaluation)

SECONDARY OUTCOMES:
Number of adverse events | 0-6 weeks
  Number of adverse events (total and per causality category)
Change in stool consistency | Change from week 0 to week 4
  Change in stool consistency according to Bristol stool form scale (subjective evaluation; range from Type 1 as separate hard lumps to Type 7 as liquid consistency with no solid pieces)
Change in defecation frequency | Change from week 0 to week 4
  Change in defecation frequency according to visual analogue scale (VAS; score 0-100; subjective outcome)
Change in clinical significance status of screening blood safety tests | Change from week -2 to week 4
  Change in clinical significance status of screening blood safety tests
Change in body mass index (BMI) | Change from week -2 to week 4
  Change in BMI due to weight change
Palatability | 2-4 weeks
  Palatability of investigational product according to visual analogue scale (VAS; score 0-100; subjective outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Nieminen, MD, Principal Investigator — Satucon Oy
Locations (1):
- Satucon Oy/Pihlajalinna Ite, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No